CLINICAL TRIAL: NCT04314310
Title: Effects on Recovery of Postoperative Gastrointestinal Function With Multimodal Analgesia in Patients Receiving Abdominal and Non-abdominal Surgeries.
Brief Title: Effects on Recovery of Postoperative Gastrointestinal Function With Multimodal Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201912245RINB
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Recovery
Keywords: orocecal transmit time, flatus
MeSH Terms: conditions — Flatulence | interventions — tenoxicam

STUDY DESIGN:
Intervention Model Description: treatment: Tenoxicam; control: placebo
Who Masked: Participant, Care Provider
Masking Description: care provider and participant were masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenoxicam (Active Comparator): nonsteroidal anti-inflammatory drug (NSAID)
  Interventions: Drug: Tenoxicam
- placebo (Placebo Comparator): equal volume of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenoxicam — nonsteroidal anti-inflammatory drug (NSAID)
  Arms: Tenoxicam
Drug: Placebo — equal volume of normal saline
  Arms: placebo

SUMMARY:
breast cancer surgery is associated with a high incidence of persistant postsurgical pain (PPSP). The aim of the study was to evluate the impact of intravenous Tenoxicam on acute and PPSP, analgesic requirements and gastrointestinal recovery in patients undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
thrity patients participated in this randomized, single-blined study. Before and at the postoperative day 1, the bowel function (orocecal transmit time) were measured. Before induction of general anesthesia, patients recieved a bolus of intravenous Tenoxicam or an equal volume of saline (control group). Pain score and opioid consumption were recorded in the postoperative period and then daily for 1 week.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to II Breast cancer patients Mastectomy or wide local excision + axillary note dissection

Exclusion Criteria:

* Preexisting malignancy Chronic infection Previous pain condition Diabetes Thyroid disorder Severe cardiac, renal or hepatic disease Previous breast surgery Psychiatric illness Neurological disease Contraindication for tenoxicam or morphine use

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-23 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | until postoperative day7
  morphine consumption after breast cancer surgery

SECONDARY OUTCOMES:
orocecal transmit time, | preoperative and postoperative day 1
  smal intestinal function

IPD SHARING:
Plan to Share IPD: No
due to ethical concern